CLINICAL TRIAL: NCT05503498
Title: Population Pharmacokinetic Modeling of Fibrinogen in Patients With Congenital or Acquired -Chronic or Acute- Hypofibrinogenemia
Brief Title: Pharmacokinetic Model of Fibrinogen Plasma Levels After Fibrinogen Administration
Acronym: PKMF
Status: Completed | Type: Observational
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: University of Barcelona (Other)
Responsible Party: Principal Investigator, Annabel Blasi, principal investigator, Hospital Clinic of Barcelona
Other Study IDs: PMODEL
Record Dates: First submitted 2022-08-11; First posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Fibrinogen; Deficiency, Acquired; PHARMACOKINETICS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AFIBRINOGENEMIA, CIRRHOSIS, TRAUMATICS: PATIENTS WITH CONGENIAL AFIBRINOGENEMIA:RECORD OF PLASMA FIBRINOGEN LEVEL PATIENTS WITH ADQUIRED CRONIC HIPOFIBRINOGENEMIA AND END STAGE OF THE LIVER DISEASE: RECORD OF PLASMA FIBRINOGEN LEVEL PATIENTS WITH ADQUIRED ACUTE HIPOFIBRINOGENEMIA AND ACUTE TRAUMA: RECORD OF PLASMA FIBRINOGEN LEVEL
  Interventions: Other: DATA RECORDING

INTERVENTIONS:
Other: DATA RECORDING — RECORD PLASMA FIBRI LEVELS AFTER FIBRINOGEN ADMINISTRATION

SUMMARY:
characterize the fibrinogen PK in patients with acquired -chronic (cirrhotic patients) or acute- hypofibrinogenemia (severe trauma or critical haermorrhage), showing endogenous production.

DETAILED DESCRIPTION:
Fibrinogen, a plasma-soluble protein synthesized by the liver, is the key substrate for the plasmatic blood coagulation, reaching a critically low plasma concentration earlier than other coagulation factors in case of bleeding. Fibrinogen Pharmacokinetics (PK) after single doses of fibrinogen concentrate (FC), using modeling approaches, has only been evaluated in congenital afibrinogenaemic patients. The aims of this study are to extend the modeling process to characterize the fibrinogen PK in patients with acquired -chronic (cirrhotic patients) or acute- hypofibrinogenemia (severe trauma or critical haermorrhage), showing endogenous production. Influencing factors of differences on the fibrinogen PK between sub-populations will be identified.

ELIGIBILITY:
Inclusion Criteria: AFIBRINOGENEMIC, TRAUMATIC AND CIRRHOTIC AFTER FIBRINOGEN ADMINISTRATION -

Exclusion Criteria: NA

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: AFIBRINOGENEMIC, TRAUMATIC AND CIRRHOTIC AFTER FIBRINOGEN ADMINISTRATION
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
plasma fibrinogen level | JUNE 2021- AUGUST 2022
  to develop a pharmacokinetic model to predict the plasma fibrinogen level after fibrinogen administration

CONTACTS AND LOCATIONS:
Overall Officials: ANNABEL NA BLASI, PMPHD, Principal Investigator — Hospital Clinic of Barcelona
Locations (2):
- Spain (2):
  - Hospital Clinic, Barcelona
  - Hospitla Clinic, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided
PUBLICATION